CLINICAL TRIAL: NCT01092065
Title: A 6-week, Double-blind, Placebo-controlled, Randomized, Multicenter Study to Explore the Efficacy and Safety of AFQ056 When Combined With Increased Doses of L-dopa in Parkinson's Disease Patients With OFF Time and Moderate-severe L-dopa Induced Dyskinesia
Brief Title: Efficacy and Safety of AFQ056 When Combined With Increased Doses of L-dopa in Parkinson's Disease Patients With Moderate-severe L-dopa Induced Dyskinesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAFQ056A2216
Record Dates: First submitted 2010-03-22; First posted 2010-03-24 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2013-03

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Dyskinesia; Drug-induced; Levodopa; L-dopa
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — mavoglurant; Levodopa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- AFQ056 100 mg (Bid) (Experimental)
  Interventions: Drug: AFQ056 with L-dopa
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AFQ056 with L-dopa — hard gelatin capsule to be taken bid for six weeks
  Arms: AFQ056 100 mg (Bid)
Drug: Placebo — hard gelatin capsule to be taken bid for six weeks
  Arms: Placebo

SUMMARY:
This Phase IIb exploratory study is designed to determine whether AFQ056 is safe and effective and whether it can increase the therapeutic window of L-dopa in patients whose control of their Parkinson's Disease symptoms is limited by the development of dyskinesia induced by use of L-dopa.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with Parkinson's Disease (PD), treated with L-dopa, experiencing OFF time and dyskinesias for at least three months

Exclusion Criteria:

* Surgical treatment for PD
* Cancer within the past 5 years (other than localized skin cancer and prostate cancer that has been effectively treated)
* Advanced, severe or unstable disease (other than PD) that may interfere with the study outcome evaluations

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline to the last-observation-carried-forward (LOCF) endpoint at week 5 in total OFF time collected from the Hauser et al. patient diary | 5 weeks

SECONDARY OUTCOMES:
Change from baseline to the LOCF endpoint at week 5 in ON time with dyskinesia collected from the Hauser et al. patient diary. | 5 weeks
Effect of increasing L-dopa doses on the underlying symptoms of Parkinson's Disease (PD) as measured by the United Parkinson's Disease Rating Scale (UPDRS) Part III. | 5 weeks
Change in dyskinesia from baseline to the LOCF endpoint at week 5 as measured by the modified Abnormal Involuntary Movement Scale (AIMS), patient diary and Unified Dyskinesia Rating Scale (UDysRS) Parts I-IV. | 5 weeks
Change from baseline on patient's dyskinesia, disability caused by dyskinesia and the underlying symptoms of PD as assessed by a clinician-rated (CGIC) and a patient-rated (PGIC) global impression of change. | 5 weeks
Safety and tolerability as measured by changes in vital signs, laboratory values, ECGs, and percentages of treatment-emergent AEs and SAEs | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (4):
  - The Parkinsons Institute, Sunnyvale, California
  - Colorado Neurological Institute, Englewood, Colorado
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Kansas Medical Center - Parkinson's Disease and Movement Disorders Center, Kansas City, Kansas

REFERENCES:
- See also: Results for CAFQ056A2216 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=6483